CLINICAL TRIAL: NCT01030042
Title: Randomized, Phase III, Multicenter Trial Comparing Two Different Sequences of therapyFOLFOX-4 vs FOLFOX-4 Followed by Irinotecan/Cetuximab in Metastatic Colorectal Patients Treated With FOLFIRI /Bevacizumab as First Line Chemotherapy
Brief Title: Trial Comparing Two Two Sequences of Therapy in Colorectal Metastatic Patients
Acronym: COMETS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-006254-26
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2009-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic; colorectal cancer; two sequences therapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Folfox protocol; Oxaliplatin; Fluorouracil; Leucovorin; Irinotecan; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cetuximab/Irinotecan (Experimental): Cetuximab/irinotecan followed, after progression, by FOLFOX-4 (Oxaliplatin, leucovorin and 5-fluorouracil)
  Interventions: Drug: Irinotecan/Cetuximab
- FOLFOX 4 (Active Comparator): FOLFOX-4 (Oxaliplatin, leucovorin and 5-fluorouracil) followed, after progression, by irinotecan/cetuximab
  Interventions: Drug: FOLFOX-4

INTERVENTIONS:
Drug: FOLFOX-4 — Day 1: OXA will be administered as a 85 mg/m2 iv infusion over 2 hours; Leucovorin as a 100 mg/m2 infusion over 2 hours, 5-FU will be given as a 400 mg/m2 bolus injection, and then as a 600 mg/m2 continuous infusion over 22 hours after the first infusion Day 2: Leucovorin 100 mg/m2 (alone), followed by 5-FU 400 mg/m2 bolus injection, and 5-FU 600 mg/m2 continuous infusion after the first infusion Cycle length is 2 weeks comprising approximately 48 hours of infusion and 12 days of rest. Cycles are to be repeated every second week for a total of either 6 (12 weeks) or 12 cycles (24 weeks).
  Other Names: Oxaliplatin, 5FU, Leucovorin
  Arms: FOLFOX 4
Drug: Irinotecan/Cetuximab — CET 400 mg/m2 intravenously via infusion pump given over a 120 min time and weekly CET infusions at a maintenance dose of 250 mg/m2 given over a 60 min time.
  IRI 180 mg/m2 iv infusion over 30-90 min. Cycle length is 2 weeks and it is to be repeated until disease progression.
  Other Names: CPT11/Cetuximab
  Arms: Cetuximab/Irinotecan

SUMMARY:
Primary Objectives:

Aim of this study is to compare the efficacy and safety of two different sequences of chemotherapeutic agents in order to optimize the treatment of patients with metastatic colorectal cancer progressed to a first line chemotherapy with FOLFIRI and bevacizumab. Primary endpoint will be overall survival, defined as the time elapsed from the date of randomization to the date of patient death due to any cause, or the last date the patient was known to be alive.

Secondary Objectives Progression free survival, Quality of life, Health resource utilisation and economic evaluation, Toxicity and incidence of adverse events

The study regimen includes:

Strategy A: FOLFOX-4 followed, after progression, by irinotecan/cetuximab Strategy B: irinotecan/cetuximab followed, after progression, by FOLFOX-4 Patients will be randomly assigned to one of the two treatment sequences (with 1:1 ratio) using a block design randomization procedure stratified according to center.

The patient accrual period is planned for approximately 36 months. To assess OS, all pts will be followed for up to 18 months after the last patient is randomised. The maximum estimated study duration is approximately 54 months.All statistical analyses will be based on an intention-to-treat approach. CONSORT rules will be applied to describe study flow and protocol deviations.

DETAILED DESCRIPTION:
Target population:

Patients with histologically confirmed metastatic colorectal cancer progressed after a first line treatment containing FOLFIRI and BEV

Inclusion criteria:

* Age >18 < 75 years of age
* Diagnosis of histologically proven adenocarcinoma of the colon or rectum, stage IV
* K-ras wild-type
* ECOG performance status 0-1 at study entry

Endpoints:

- Response Rate, Disease control rate, The duration of overall response, Overall survival, PFS, Time to treatment failure, Quality of Life, Incidence of AEs, Frequency and nature of serious adverse reactions (SADRs), Premature withdrawals

Statistical methods:

Assuming a randomization ratio of 1:1, 282 deaths are required in order to achieve a power of 80% of detecting a hazard ratio of 0.72 in favour of one of the two sequences, translating in an increase of median survival time from 10 to 14 months, with a type I error of 5%, two-sided, using the Mantel-Cox version of the log-rank test. With a uniform accrual period of 3 years and a follow-up of 18 months, about 350 patients will be needed to reach the target number of events.

All statistical analyses will be based on an intention-to-treat approach. CONSORT rules will be applied to describe study flow and protocol deviations.

All OS and PFS curves will be drawn with the Kaplan-Meier method. Results will be presented as Hazard Ratio (HRs) and their 95% Confidence Interval (CIs).

On annual basis, starting from the second year, an interim analysis will be conducted. In principle, no formal stopping rule will be applied, unless otherwise suggested by the DSMC. Safety reports will be drawn on annual basis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 <75 years of age
* Diagnosis of histologically proven adenocarcinoma of the colon or rectum, stage IV
* K-ras wild-type
* Performance Status (ECOG-PS) 0-1 at study entry
* Neutrophils ≥ 1.5 x 1039/L, platelets ≥ 100 x 109/L, and hemoglobin ≥ 9 g/dL
* Bilirubin level either normal or < 1.5 x upper limit of normal (ULN)
* Asparagine aminotransferase (ASAT) and alanine aminotransferase (ALAT) ≤ 2.5 X ULN (≤ 5 x ULN if liver metastasis are present)
* Serum creatinine < 1.5 x ULN
* Effective contraception for both male and female patients
* Life expectancy of ≥ 3 months
* Signed written informed consent

Exclusion Criteria:

* History or presence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or patient at high risk from treatment complications
* Other malignancies within the last 5 years (other than curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix)
* History of psychiatric disability judged by the investigator to be clinically significant, precluding informed consent or interfering with compliance for oral drug intake
* Known grade 3 or 4 allergic reaction to any of the components of the treatment
* Known drug abuse/ alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-09; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Overall Survival | the time from the date of randomisation to the date of death

SECONDARY OUTCOMES:
Progression free survival | the time relapsed from the date of randomization and the date of progression after third-line treatment or death

CONTACTS AND LOCATIONS:
Locations (32):
- Italy (32):
  - A.O. Ospedale Umberto I - Università - Località Torretta, Ancona, Ancona
  - Ospedale Profili, Fabriano, AN
  - Usl 11 Ospedale Murri, Fermo, AP
  - Ospedali Riuniti, Largo Barozzi, 1, Bergamo, Bergamo
  - A.O. Treviglio-Caravaggio, P.le Ospedale n1, Treviglio, Bergamo
  - Fondazione Poliambulanza, Via Bissolati 57, Brescia, Brescia
  - Spedali Civili, Brescia, BS
  - AUSL di Lanciano-Vasto, Lanciano, CH
  - Istituto Oncologico del Mediterraneo, Catania, CT
  - ASL 11, Empoli, FI
  - Università, Florence, FI
  - A.O. Ospedale S.Anna, Como, Italy
  - Ospedale Maggiore, Lodi, LO
  - A.O. Carlo Poma - Via Albertoni, 1, Mantova, Mantova
  - Ospedale S.Vincenzo, Taormina, ME
  - Ospedale Serbelloni, Gorgonzola, MI
  - Istituto di Ricerca S.Raffaele, Milan, MI
  - Ospedale Fatebenefratelli, Milan, MI
  - A.O. S.Gerardo, Monza, MI
  - Istituto Oncologico Veneto, Padua, PD
  - A.O. S.Salvatore, Pesaro, PS
  - Ospedale Civile, Urbino, PS
  - Azienda Ospedaliera San Carlo, Potenza, PZ
  - Università Policlinico Umberto I, Roma, RM
  - Ospedale Sant'Andrea, Roma, RM
  - Università Campus Biomedico, Via Emilio Longoni, 83, Roma, Roma
  - A.O. S.Giovanni Calabita Fatebenefratelli, Roma, Roma
  - AULSS 18 di Rovigo, Rovigo, RO
  - Ospedale Morelli, Sondalo, SO
  - Università degli Studi, Candiolo, TO
  - Ospedale Mater Salutis, Legnago, VR
  - Istituto Tumori - Fondazione Pascale, Napoli